CLINICAL TRIAL: NCT06059742
Title: The Effects of Action Observation Therapy With and Without Acoustic Stimulation on Balance and Gait Among Stroke Survivors
Brief Title: Action Observation Therapy With and Without Acoustic Stimulation in Post Stroke Gait and Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS-ISB/REC/01642
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy with Acoustic Stimulation (Experimental): The patients in the action observation therapy with acoustic stimulation group will be required to observe the lower limb movements or functional actions with sound of beats in video clips. (i.e., the observation phase) and to execute what they had observed to the best of their ability with sound of beats given through headphones (i.e., the execution phase). Three common categories of movements will be elected in the protocol for each week based on the related literature
  Interventions: Other: Action Observation Therapy with Rhythmic acoustic stimulation
- Action Observation Therapy Without Acoustic Stimulation (Active Comparator): The patients in the action observation therapy without acoustic stimulation group will be required to observe the lower limb movements or functional actions without sound of beats in video clips. (i.e., the observation phase) and to execute what they had observed to the best of their ability without sound of beats (i.e., the execution phase). Three common categories of movements will be elected in the protocol for each week based on the related literature
  Interventions: Other: Action Observation Therapy without Rhythmic acoustic stimulation

INTERVENTIONS:
Other: Action Observation Therapy with Rhythmic acoustic stimulation — Action observation therapy is observing some action and the performing Rhythmic acoustic stimulation is performing movement on the rhythm of beats
  Arms: Action Observation Therapy with Acoustic Stimulation
Other: Action Observation Therapy without Rhythmic acoustic stimulation — Action observation therapy is observing some action and the performing Rhythmic acoustic stimulation is performing movement on the rhythm of beats
  Arms: Action Observation Therapy Without Acoustic Stimulation

SUMMARY:
Stroke causes the interruption of blood flow towards the brain cells which results in cell death and lead to variety of disorders including deficits in balance and gait. It is well known that it is causing death and disability .The incidence of stroke is increasing in low-income countries because of not using evidence-based practice in health-related conditions in these countries. Action observation training is one of the new developing rehabilitation technique that targets motor learning by the activation of mirror neurons and is the most important approach that targets the motor and functional recovery in stroke patients. A new treatment approach i .e action observation therapy, in which the movements are observed by the patient to provide visual stimulus, then patients are asked to perform those movements. A new approach acoustic stimulation is introduced for improving gait and balance in post stroke patients in which individual patient cadence is used to adjust the beats of sound so that auditory stimulation causes recovery.

DETAILED DESCRIPTION:
Stroke is a medical condition which causes the cessation of blood flow to the brain cells and results in cell death. It is a leading cause of death and disability. Geographical variations play a huge role in the burden for stroke. A stroke survivor experiences a range of symptoms that make it harder for them to carry out regular tasks and raise their risk of falling while walking .The effects of Action Observation Therapy with acoustic stimulation on balance in stroke patients have not been explicitly covered in recent studies. The study intends to evaluate the effectiveness of treatments with evidence for post-stroke balance and gait.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Both male and female
* Any type of stroke
* Walking few steps [5 or more] .
* Berg balance score above 21
* Ability to follow the study instructions-Mini mental state examination (MMSE ) score >24

Exclusion Criteria:

* Patients diagnosed with other neurological diseases
* Tumors or neoplasms
* Cardiopulmonary diseases
* Patient with impaired cognition
* Visual and auditory impairments

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | week 8
  It is often used to assess balance and mobility as well as identify people who are at risk of falling. 14 different balance-related tasks, including sitting, standing, and transferring, are included in the tool. Each factor is scored from 0 to 4, with 0 suggesting significant impairment and 4 denoting the patient's balance system operating normally
Wisconsin Gait Scale | week 8
  Wisconsin Gait Scale is an observational tool for the evaluation of gait quality in individuals after stroke with hemiplegia. It is divided into four sub scales, which assess a total of fourteen spatiotemporal and kinematic parameters of gait observed during the consecutive gait phases.
Time Up and Go Test | week 8
  The Timed Up and Go test, which integrates elements of gait and balance control, has primarily been used to predict the risk of falling in geriatric populations. Patients are instructed to stand up from a chair, move 3 meters at a safe and comfortable speed, turn around, and then return to the chair and sit down.
6 Min Walk Test | week 8
  it is a simple and effective test that requires the subject to walk as fast as they can for six minutes. Because of this, it relies on patient-determined, individually modified parameters, and patients are even permitted to quit walking if they so desire

SECONDARY OUTCOMES:
Functional Reach Test | week 8
  A static balance test called the functional reach test is frequently used to evaluate a subject's level of balance when they are standing.The reach distance during this has been used as a measurement for determining fall risk

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD*, Principal Investigator — Riphah International University
Locations (1):
- HBS hospital Lehtrar Road Alipur, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No